CLINICAL TRIAL: NCT05517434
Title: Intra-Articular Autologous Bone Marrow Aspirate vs Placebo Injection and Lipoaspirate Micronized With Leukocyte-Poor Platelet Rich Plasma vs Placebo Injection Evaluations for Treatment of Knee OsteoArthritis: The ABLE OA Double-Blinded Randomized Clinical Trial
Brief Title: Autologous BMA vs Saline and LAM + LP-PRP vs Saline Evaluations in Knee OA
Acronym: ABLE-OA
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-5959; 22-5792 (ABLE OA, study 2) (Other: University Health Network)
Record Dates: First submitted 2022-08-19; First posted 2022-08-26 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis, Knee
Keywords: placebo; intra-articular injection; autologous therapy; bone marrow aspirate; lipoaspirate; platelet-rich plasma; leukocyte-poor; pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Sodium Chloride; cyclomaltodextrin glucanotransferase; lipoarabinomannan

STUDY DESIGN:
Intervention Model Description: STUDY 1 (N=74): All patients will undergo a bone marrow aspiration. A BMA injection [Arm A, n=37] will be compared to a saline injection [Arm C, n=37].
  STUDY 2 (N=74): All patients will undergo a blood collection and lipoaspiration. A LAM injection followed by LP-PRP injection [Arm B, n=37] will be compared to two consecutive saline injections [Arm D, n=37].
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A research nurse/staff will prepare the minimally manipulated cellular preparations and injection syringe(s), as well as deliver the corresponding syringe(s) based on group allocation to the clinician to administer the injection into the patient's knee joint. The syringe(s) containing the active treatment or saline solution will be obscured by a non-transparent, adhesive label hiding its content in order to maintain the blind for both the patient and clinician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- For STUDY 1 (ARM A): Bone Marrow Aspirate (BMA) (Experimental): This group will undergo a bone marrow aspiration and receive an ultrasound guided intra-articular injection of BMA (a single dose of cellular suspension of 9 mL or less)
  Interventions: Biological: Bone Marrow Aspirate (BMA): Minimally manipulated autologous cellular preparation
- For STUDY 1 (ARM C): Saline Injection (Placebo Comparator): This group will undergo a bone marrow aspiration and receive an ultrasound guided intra-articular injection of saline solution (9 mL)
  Interventions: Other: Saline (Placebo Comparator for BMA)
- For STUDY 2 (ARM B): Lipoaspirate Micronized + Leukocyte-Poor Platelet-Rich Plasma (LAM + LP-PRP) (Experimental): This group will undergo a blood collection plus lipoaspiration and receive an ultrasound guided intra-articular injection of LAM (a single dose of cellular suspension of 9 mL or less) followed by LP-PRP (a single dose of cellular suspension of 2 mL or less)
  Interventions: Biological: Lipoaspirate Micronized + Leukocyte-Poor Platelet-Rich Plasma (LAM + LP-PRP): Minimally manipulated autologous cellular preparations
- For STUDY 2 (ARM D): Saline Injection (Placebo Comparator): This group will undergo a blood collection plus lipoaspiration and receive ultrasound guided intra-articular injections of saline solution (9 mL followed by 2 mL)
  Interventions: Other: Saline (Placebo Comparator for LAM + LP-PRP)

INTERVENTIONS:
Biological: Bone Marrow Aspirate (BMA): Minimally manipulated autologous cellular preparation — Participants will undergo a bone marrow aspiration. About 10 mL of BMA will be collected from the posterior iliac spine i.e., ipsilateral and/or contralateral iliac crest using the Cervos Marrow Cellution™ kit. The BMA does not require processing using a centrifuge after collection. 9 mL (or less) of BMA is injected into the osteoarthritic knee joint after collection (Arm A, Study 1).
  Arms: For STUDY 1 (ARM A): Bone Marrow Aspirate (BMA)
Other: Saline (Placebo Comparator for BMA) — Participants will undergo a bone marrow aspiration to collect about 10 mL of BMA from the posterior iliac spine i.e., ipsilateral and/or contralateral iliac crest. However, 0.9% sodium chloride (NaCl) Baxter or equivalent (9 mL) is injected into the osteoarthritic knee joint (Arm C, Study 1).
  Arms: For STUDY 1 (ARM C): Saline Injection
Biological: Lipoaspirate Micronized + Leukocyte-Poor Platelet-Rich Plasma (LAM + LP-PRP): Minimally manipulated autologous cellular preparations — Participants will undergo a lipoaspiration. 40 mL of lipoaspirate (LA) will be collected from subcutaneous adipose tissue. LA will be processed using the Cervos LIPO-PRO™ kit and a centrifuge. Participants will also undergo a blood draw. About 30 mL of whole blood will be collected from the antecubital fossa. Whole blood will be processed using the Cervos KEYPRP kit and a centrifuge. After processing, 9 mL (or less) of LAM is injected first followed immediately by 2 mL (or less) of LP-PRP into the osteoarthritic knee joint (Arm B, Study 2).
  Arms: For STUDY 2 (ARM B): Lipoaspirate Micronized + Leukocyte-Poor Platelet-Rich Plasma (LAM + LP-PRP)
Other: Saline (Placebo Comparator for LAM + LP-PRP) — Participants will undergo a lipoaspiration to collect 40 mL of LA and a blood draw to collect about 30 mL of whole blood. However, 0.9% of sodium chloride (NaCl) Baxter or equivalent is injected twice (9 mL + 2 mL) into the osteoarthritic knee joint (Arm D, Study 2).
  Arms: For STUDY 2 (ARM D): Saline Injection

SUMMARY:
ABLE OA is a Health Canada authorized (phase II/III) trial [Parent Control #: 263591]. A multi-center, prospective, double-blinded, randomized, placebo-controlled adaptive trial to evaluate the efficacy of two minimally manipulated autologous cellular preparations i) bone marrow aspirate (BMA) injection; and, ii) combined lipoaspirate micronized (LAM) and leukocyte poor (LP) platelet-rich plasma (PRP) injections for the treatment of knee osteoarthritis (OA).

BMA, LAM from lipoaspirate (LA), and LP-PRP from whole blood will be prepared using the Cervos Marrow Cellution™ Bone Marrow Aspiration System, Cervos LIPO-PRO™ Adipose Transfer System, and Cervos KEYPRP Platelet Separator System, respectively.

Patient-reported outcome (PRO) measures will be collected using web- or paper-based questionnaires administered at baseline (pre-injection) as well as at 3, 6 and 12 months (post-injection). Blood, synovial fluid, and urine samples will be collected at baseline pre-injection and 6 months post-injection only.

DETAILED DESCRIPTION:
Trial interventions will occur in two independent studies under a single protocol where each experimental treatment will be compared to a placebo control.

Our primary hypothesis is that BMA or LAM + LP-PRP injection is 35% more effective than placebo saline injection control in terms of response rates in Numeric Pain Rating Scale (NPRS) scores as measured by their difference.

PRIMARY OBJECTIVE:

To determine the efficacy of an intra-articular injection of BMA or LAM + LP-PRP in patients with knee OA by comparing each of the two treatments to a placebo saline injection control arm. Efficacy will be measured by a pain intensity improvement of a minimum of 2 points in NPRS scores at 6 months after injection relative to baseline. The study endpoint is 6 months post-injection.

KEY SECONDARY OBJECTIVE:

To determine efficacy measured by improvements in the Knee Injury and Osteoarthritis Outcome Score (KOOS) function activities of daily living (ADL) subscale scores at 6 months after injection relative to baseline by comparing each of the treatment (BMA or LAM + LP-PRP) arm to a placebo saline control arm.

OTHER SECONDARY OBJECTIVES:

* To evaluate if an injection of BMA or LAM + LP-PRP into the knee joint shows greater improvements in other pain outcomes (including KOOS pain) compared to placebo injection at 3, 6 and 12 months post-injection relative to baseline.
* To evaluate the safety of BMA or LAM + LP-PRP injection into the knee joint compared to placebo injection. Adverse events will be collected at baseline, 3, 6 and 12 months post-injection, and deleterious effects on the joint will be assessed by X-ray at 6 months post-injection only.
* To evaluate the health profile and overall self-rated health status of patients in treatment and placebo arms at 3, 6 and 12 months post-injection relative to baseline.
* To evaluate overall patient satisfaction in treatment and placebo arms at 6 months post-injection.
* To evaluate health care consumption and health-related productivity losses of paid and unpaid work using the iMTA Medical Consumption Questionnaire (iMCQ) and iMTA Productivity Cost Questionnaire (iPCQ), respectively at 6 and 12 months post-injection relative to baseline.
* To determine the quality-adjusted-life years (QALYs) using the 5-level EuroQol five-dimensional (EQ-5D-5L) health state utility scores based on the Canadian preference weights to inform cost-effective estimates.

EXPLORATORY OBJECTIVES:

To determine the correlation between changes in NPRS/KOOS pain scores and KOOS ADL function at 6 months relative to baseline and the heterogeneity in:

1. the cellular composition and soluble factors in BMA, LAM and LP-PRP autologous cellular preparations [in BMA or LAM + LP-PRP groups only]
2. the levels of local and systemic immune cell and inflammatory profiles of patients (based on synovial fluid, blood, and urine readouts) [in BMA or LAM + LP-PRP and placebo groups]

A total of approximately 84 eligible participants in each study will be randomized in a 1:1 ratio, which allows for 42 participants per group (treatment vs. placebo). This sample size considers a potential drop-out rate of 10% for each study. Three recruitment centres (Toronto Western Hospital (TWH), University Health Network (UHN); Women's College Hospital (WCH); Cleveland Clinic Canada (CCC)) and one treatment centre (TWH, UHN) will be involved in these two studies. Stratification will occur by centre, baseline NPRS of 4-6 (moderate pain) or 7-10 (severe pain), and KL grade of 2 (minimal OA) or 3 (moderate OA). Additionally, the need to re-estimate the required sample size will be evaluated using the information available at interim. At the interim analysis, contingent on observed response rates and corresponding statistical signal, the required sample size may increase, ranging from 100 to 288 patients in total for each of the two studies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 30 years of age at the time of screening
* Willingness and ability to comply with study procedures and visit schedules and able to follow oral and written instructions
* Signed consent for study participation
* Baseline NPRS ≥ 4 points
* Presence of chronic, symptomatic knee pain in at least one knee; if both knees are affected, the knee with greater severity will be selected for treatment
* KL grade 2 or 3 knee OA based on standing knee X-ray assessment
* Body mass index ≤ 30 kg/m2

Exclusion Criteria:

* Approved anti-inflammatory therapy injections (corticosteroid, Synvisc, PRP, nSTRIDE-Autologous Protein Solution) within the previous 6 months in the knee
* Major axial deviation (varus >10°, valgus >10°)
* Any concomitant knee lesion causing pain or effusion (i.e., ligamentous or meniscal injury, osteochondral lesion)
* Presence of clinically observed active infection in the index knee
* Diagnosed with rheumatoid arthritis, Reiter's syndrome, psoriatic arthritis, gout, ankylosing spondylitis, or arthritis secondary to other inflammatory diseases; chondrocalcinosis, Paget's disease, or villonodular synovitis
* Diagnosed with leukemia or other hematologic cancers, known presence of metastatic malignant cells, or ongoing or planned chemotherapeutic treatment
* Presence of venous or lymphatic stasis in the index leg
* A history of local anesthetic allergy
* Medical conditions such as hemophilia or other blood clotting disorders
* Arthroscopic knee surgery within the previous 6 months
* Daily opioid use for the past 3 months, use of non-steroidal anti-inflammatory drugs within 1 week of the procedure, unable to hold anti-platelet medications
* Use of systemic corticosteroids for treatment of a chronic medical condition within the past 3 months
* Immunosuppression or acute infective processes

Study Treatment Exclusion:

* For Study 1: Inability to tolerate the bone marrow aspiration procedure resulting in insufficient collection of BMA (<10 mL) after two successive aspiration attempts
* For Study 2: Inability to tolerate the lipoaspiration procedure resulting in insufficient collection of LA (<40 mL) after two successive aspiration attempts

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain Level Changes. Differences in response rates between groups (treatments vs placebos) at 6-months (end of study) compared to baseline. Response is based on an improvement of 2 units or more in the Numeric Pain Rating Scale (NPRS). | baseline (pre-injection) and 3, 6 and 12 months (post-injection)
  Pain intensity will be measured by the NPRS. The score ranges from 0 to 10, with 0 indicating "No Pain" and 10 "Worst Imaginable Pain".

SECONDARY OUTCOMES:
Functional Changes. Differences in mean change of Knee Injury and Osteoarthritis Outcome Score (KOOS) Activities of Daily Living (ADL) subscale scores between groups (treatments vs placebos) at 6-months (end of study) compared to baseline. | baseline (pre-injection) and 3, 6 and 12 months (post-injection)
  KOOS was originally developed in 1995 by Ewa M Roos and colleagues. The KOOS was developed as an extension of the WOMAC Osteoarthritis Index with the purpose of evaluating short- and long-term symptoms and function in subjects with knee injury and OA. It holds 42 items in 5 separately scored subscales: Pain, other Symptoms, Function in Daily Living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL). Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Additional Pain Level Changes. Mean NPRS subscale change score at 6 months relative to baseline in treatment groups compared to placebo groups. | baseline (pre-injection) and 3, 6 and 12 months (post-injection)
  See above for description of NPRS.
Additional Pain Level Changes. Mean KOOS pain subscale change score at 6 months relative to baseline in treatment groups compared to placebo groups. | baseline (pre-injection) and 3, 6 and 12 months (post-injection)
  See above for description of KOOS.
Health-Related Quality of Life Changes. Mean utility and EuroQol-Visual Analogue Scale (EQ-VAS) change scores at 6 months (end of study) relative to baseline in treatment groups compared to placebo groups. | baseline (pre-injection) and 3, 6 and 12 months (post-injection)
  EQ-5D-5L is a commonly used generic preference-based health-related QOL measure. It is a multi-attribute instrument, which considers five dimensions including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Respondents are asked to rate their health today on each dimension. Each dimension has five levels of severity i.e., no problems (level 1); slight; moderate; severe; and extreme problems (level 5). There are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health). The health states are converted into a single index 'utility' score using a scoring algorithm. There is also a VAS, which is used as a quantitative measure of overall health status i.e., 0 represents the worst health you can imagine and 100 represents the best health you can imagine.
Safety. Proportion of cumulative adverse events (AEs) at 6 months post-injection in treatment groups compared to placebo groups. | baseline (pre-injection) and 3, 6 and 12 months (post-injection)
  AEs will either be sought by the clinician via non-directive questioning, by clinical exam at scheduled visits, and/or detected when volunteered by the study participant during or between visits. At the 6-month visit, deleterious effects on the joint will also be assessed by X-ray of the knee. AEs beyond the 6-month visit will be addressed according to standard clinical management practices. A statement that a patient had no AEs also constitutes a safety assessment.
Treatment Satisfaction. Percent satisfaction at 6 months in treatment groups compared to placebo groups. | 6 months (post-injection)
  This will be evaluated with a single question with five response options (very dissatisfied; somewhat dissatisfied; neither dissatisfied or satisfied; somewhat satisfied; very satisfied).

OTHER OUTCOMES:
Total nucleated cell count (TNC) in the BMA and LAM cellular preparations in treatment groups only. | baseline (pre-injection) and 6 months (post-injection)
  This is to address heterogeneity in the cellular composition of cellular autologous preparations. The correlation between TNC and NPRS/KOOS pain and KOOS ADL scores at 6 months relative to baseline will be evaluated.
Percentages of hematopoietic, endothelial, and stromal cells in the BMA and LAM cellular preparations in treatment groups only. | baseline (pre-injection) and 6 months (post-injection)
  This is to address heterogeneity in the cellular composition of cellular autologous preparations. The correlation between the sub-population fractions and NPRS/KOOS pain and KOOS ADL scores at 6 months relative to baseline will be evaluated.
Levels of soluble/secreted factors (FGF2, G-CSF, IL-1RA/IL-1F3, IL-4, IL-10, PDGF-BB, VEGF) in the BMA, LAM and LP-PRP cellular preparations in treatment groups only. | baseline (pre-injection) and 6 months (post-injection)
  This is to address heterogeneity in the cellular composition of cellular autologous preparations. The correlation between soluble/secreted factor levels and NPRS/KOOS pain and KOOS ADL scores at 6 months relative to baseline will be evaluated.
Local and systemic levels of immune cells and inflammatory cytokines and chemokines in synovial fluid and blood in treatment groups and placebo groups. | baseline (pre-injection) and 6 months (post-injection)
  This is to address heterogeneity in the inflammatory/immune cell profiles of patients and evaluate correlation to NPRS/KOOS pain and KOOS ADL scores at 6 months relative to baseline.
Systemic levels of inflammatory and catabolic factors in synovial fluid, blood and urine in treatment groups and placebo groups. | baseline (pre-injection) and 6 months (post-injection)
  This is to address heterogeneity in the inflammatory/immune cell profiles of patients and evaluate correlation to NPRS/KOOS pain and KOOS ADL scores at 6 months relative to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Sowmya Viswanathan, PhD, Principal Investigator — University Health Network, Toronto; Christian Veillette, MD, MSc, FRCSC, Study Director — University Health Network, Toronto; Christopher Kim, HBSc, MSc, MD, FRCSC, PhD(c), Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Women's College Hospital, Toronto, Ontario
  - Toronto Western Hospital, University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No